CLINICAL TRIAL: NCT00193089
Title: Phase II Trial of Weekly Docetaxel, Vinorelbine, and Herceptin in the First-Line Treatment of Patients With Metastatic Breast Cancer and Overexpression of Her-2
Brief Title: Docetaxel, Vinorelbine and Trastuzumab in the Treatment of Patients With Metastatic Her-2 Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Aventis Pharmaceuticals (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 46; GIA 11180; H2369n
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Vinorelbine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Docetaxel — Docetaxel
Drug: Vinorelbine — Vinorelbine
Drug: Trastuzumab — Trastuzumab

SUMMARY:
In this phase II trial we attempt to improve upon the efficacy of the trastuzumab/vinorelbine combination by adding weekly docetaxel. When administered on a weekly schedule, docetaxel is well tolerated with minimal myelosuppression, so that it is likely that fully efficacious doses of all three drugs can be administered

DETAILED DESCRIPTION:
Upon determination of eligibility, all patients will be receive:

Trastuzumab + Vinorelbine + Docetaxel

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Metastatic breast cancer confirmed by biopsy
* Overexpression of the Her-2 oncogene
* Age > 18 years
* Measurable disease
* Able to perform activities of daily living with minimal assistance
* No previous chemotherapy for metastatic disease
* One or more previous hormonal therapies for metastatic disease.
* Adequate bone marrow, liver and kidney function
* Patients with < grade 1 peripheral neuropathy are eligible.
* Must give written informed consent prior to entering this study.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Abnormal heart function
* Previous treatment with trastuzumab
* Brain metastases untreated
* Pre-existing symptomatic peripheral neuropathy
* Serious underlying medical conditions

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2001-04; Primary Completion 2005-04 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
feasibility and toxicity of the combination of weekly docetaxel, vinorelbine, and trastuzumab in patients with metastatic breast cancer who overexpress Her-2. | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC

REFERENCES:
- [Result] Infante JR, Yardley DA, Burris HA 3rd, Greco FA, Farley CP, Webb C, Spigel DR, Hainsworth JD. Phase II trial of weekly docetaxel, vinorelbine, and trastuzumab in the first-line treatment of patients with HER2-positive metastatic breast cancer. Clin Breast Cancer. 2009 Feb;9(1):23-8. doi: 10.3816/CBC.2009.n.004. PMID 19299236